CLINICAL TRIAL: NCT01581385
Title: Acoustic Radiation Force Impulse (ARFI) Ultrasound for Noninvasive, Diagnostic Atherosclerosis Imaging; Independent Scientist: ARFI and RWI Ultrasound for Improved Atherosclerosis Imaging
Brief Title: Acoustic Radiation Force Impulse (ARFI) Ultrasound for Noninvasive, Diagnostic Atherosclerosis Imaging
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-1049; R01HL092944 (NIH)
Record Dates: First submitted 2012-03-13; First posted 2012-04-20 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; carotid artery; carotid endarterectomy
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plaque specimens extracted during clinically indicated carotid endarterectomy surgery will be sectioned and histochemically processed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: Adult patient volunteers, male and female, undergoing clinically indicated carotid endarterectomy surgery.

SUMMARY:
This is a pilot clinical trial to assess the ability of a new ultrasound-based imaging method, Acoustic Radiation Force Impulse (ARFI) ultrasound, to describe the composition and structure of atherosclerotic plaques. The hypothesis being tested is that in vivo, transcutaneous ARFI ultrasound delineates plaque composition and structure in human carotid arteries.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate Acoustic Radiation Force Impulse (ARFI) ultrasound imaging for describing the composition and structure of atherosclerotic plaques. The surgical atherosclerotic plaques of 16 patient volunteers undergoing clinically indicated carotid endarterectomy (surgical removal of plaque from the carotid artery) will be imaged preoperatively by ARFI. ARFI imaging will occur during the volunteers' preoperative workup visits (inpatient or outpatient), in the surgical holding area (inpatient or outpatient), or at the patient bedside (inpatient). Then, the routinely excised plaque specimens will be sent for histopathological processing to determine plaque composition and structure. The histopathological data will be used to validate ARFI imaging performance for plaque material and structural characterization. This will end the participant's involvement in the study.

There are two experimental components to this study beyond what is standard practice for carotid endarterectomy patients: 1) preoperative ARFI ultrasound imaging of ipsilateral (surgical) carotid arteries, and 2) submission of sections of the carotid plaque excised intraoperatively to the UNC Hospitals clinical laboratories for immunohistochemical analysis.

This study will commence with ARFI ultrasound imaging at the time of the patient volunteer's preoperative workup for carotid endarterectomy surgery (outpatients and inpatients), while the patient is in the holding area for surgery (outpatients and inpatients), or at the patient bedside (inpatients). If the patient volunteer is an outpatient, ARFI ultrasound imaging will be performed up to two weeks prior to surgery. Preoperative ARFI ultrasound imaging will be performed in addition to the patient volunteer's routine preoperative duplex ultrasound and any other exams used to determine if carotid endarterectomy is clinically indicated.

ARFI ultrasound is a noninvasive diagnostic imaging technology performed using commercially available clinical ultrasound imaging equipment - the Siemens SONOLINE or Acuson Antares imaging systems equipped for research purposes and VF10-5 or VF7-3 linear array transducers (Siemens Medical Solutions, USA Inc. Ultrasound Division). ARFI imaging will be carried out by a professional sonographer trained in peripheral vascular ultrasound and faculty (Caterina Gallippi, Ph.D., Associate Professor, study PI) and/or graduate student research assistants in the UNC-CH Joint Department of Biomedical Engineering. The sonographer will acquire ARFI ultrasound data with matched B-Mode (for anatomical reference) in ipsilateral (surgical) carotid arteries of patient volunteers. Patient volunteers will be asked to lie on an examination table (outpatients) or to remain in their hospital beds (inpatients). The head of the exam table/bed may be raised to an approximate 45 degree angle to best visualize the carotid arteries with ultrasound imaging.

Once the patient volunteer is positioned, ultrasound gel will be applied to the patient volunteer's neck. The ultrasound imaging transducer will then be placed on top of the gel. Once the carotid artery is located, ARFI ultrasound imaging will begin. In the ipsilateral (surgical) carotid artery, the imaging field of view will be centered on the carotid plaque, with axial focal depth directed to the position of the near or far wall containing the thickest portion of the plaque. Data acquisitions will be gated to diastole. Two repeated acquisitions will be acquired for each of four ARFI imaging sequences. The position of landmarks such as arterial branch points and morphological features such as arterial wall thickness will be recorded for spatial registration to duplex ultrasound and histology.

The length of time for ARFI data collection in the carotid artery is estimated to be less than 30 minutes. Once the ipsilateral (surgical) carotid artery is imaged, the study procedure will be completed for the first portion of the study.

For the second part of the study, sections of the carotid plaque specimen routinely extracted during carotid endarterectomy surgery will be photographed and then fixed and paraffin embedded in the UNC Tissue Procurement core facility. The specimens will then undergo sectioning and staining in the UNC Histopathology core facility. These experimental sections will be in addition to the sections routinely sent for immunohistochemical processing after carotid endarterectomy. Sectioning will be directed by the surgeon per standard histopathology protocol and per laboratory sampling protocol. The sections will be stained with hematoxylin and eosin (H&E) for baseline, Verhoeff van Giesen (VVG) for elastin, Sirius Red (SR) with polarized light microscopy for collagen sub-types I and III, von Kossa (VK) for calcium, and/or Lillie modification of Masson's trichrome (MT) for fibrin, or other comparable stains. This will conclude part two of the study. However, excised plaque specimens will be stored in Dr. Gallippi's (PI) laboratory for a period of up to five years following study completion. Their storage will enable re-sectioning as need to achieve proper spatial alignment with ARFI imaging. The stored specimens will not be used for future research; they are for verification purposes only. The specimens will be submerged in formalin and stored in sealed plastic containers. No identifiable information will be recorded with the samples, and all HIPAA guidelines and procedures will be observed.

Patient volunteers' participation will end once both study parts one (ARFI ultrasound imaging) and two (immunohistochemical processing of excised plaque specimens) are completed. Therefore, there will be no follow-up visits required or additional demands placed on the patient volunteers. A Patient volunteer is asked to consent to (1) ARFI ultrasound imaging of his/her ipsilateral (surgical) carotid arteries before his/her clinically indicated endarterectomy surgery, and (2) sections of his/her routinely excised plaques specimens undergoing immunohistochemical processing (in addition to any sections routinely sent for immunohistochemical processing after carotid endarterectomy). No additional procedures or requirements are proposed. Every other aspect of the volunteers' preoperative workup for surgery and the endarterectomy surgery itself will be carried out in the normal standard of care as clinically indicated.

There is no control group in this study. This is a pilot study to determine if ARFI ultrasound imaging in this patient population may be relevant to delineating the composition and structure of carotid plaques with immunohistochemical validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo clinically indicated carotid endarterectomy
* Determination of clinical need for carotid endarterectomy will be made by the vascular surgeons on this protocol, but the general criteria include symptomatic carotid disease with a stenosis or lesion in the carotid artery thought to be the source of emboli or asymptomatic carotid artery disease with a > 60% internal carotid artery stenosis in the ipsilateral (surgical) artery.
* Male or Female
* >18 years of age with no upper limit
* Ability to provide informed consent
* Surgeon's approval
* Any ethnicity or race (meeting all other criteria)

Exclusion Criteria:

* Inability to communicate in English
* Inability to provide valid consent
* Inability to remain motionless for at least 15 minutes
* Carotid arteries deeper than 35 mm
* Pregnancy*

  * Pregnant women will be excluded from this study because carotid dissection is more likely than carotid plaque in women of child-bearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years or older) male and female patients scheduled to undergo clinically indicated carotid endarterectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
ARFI AUC score | baseline
  Statistical area under the curve (AUC) scores will be calculated using trained readers and spatially matched pathologist's interpretation of histochemical data. AUC scores will be determined for each of the four ARFI beam sequences implemented in this study with respect to characterizing calcium deposits, lipid/necrotic core, fibrous caps, collagen deposits, elastin deposits, disrupted internal elastic lamina, and thrombus.

SECONDARY OUTCOMES:
ARFI sensitivity | baseline
  Statistical sensitivity will be calculated by assessing the average AUC curve across all readers for each of the four ARFI beam sequences implemented in this study with respect to characterizing calcium deposits, lipid/necrotic core, fibrous caps, collagen deposits, elastin deposits, disrupted internal elastic lamina, and thrombus.
ARFI specificity | baseline
  Statistical sensitivity will be calculated by assessing the average AUC curve across all readers for each of the four ARFI beam sequences implemented in this study with respect to characterizing calcium deposits, lipid/necrotic core, fibrous caps, collagen deposits, elastin deposits, disrupted internal elastic lamina, and thrombus.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina M Gallippi, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill Hospitals, Chapel Hill, North Carolina, United States